CLINICAL TRIAL: NCT04770220
Title: A Phase 3, Multicenter, Randomized, Double-blind, Placebo-controlled Study of the Efficacy, Safety and Biomarker Effects of ALZ-801 in Subjects With Early Alzheimer's Disease and APOE4/4 Genotype
Brief Title: An Efficacy and Safety Study of ALZ-801 in APOE4/4 Early AD Subjects
Acronym: APOLLOE4
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alzheon Inc. (Industry)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ALZ-801-AD301; R01AG065253 (NIH); 2020-005755-20 (EudraCT Number)
Record Dates: First submitted 2021-02-22; First posted 2021-02-25 (Actual); Results first posted 2025-11-10 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-10

CONDITIONS: Early Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Intervention Model Description: This is a multi-center Phase 3, randomized, double-blind, placebo-controlled, parallel-group study.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ALZ-801 (Experimental): ALZ-801 265 mg BID tablet orally. Subjects will receive placebo in the morning and one tablet of ALZ-801 265 mg tablet in the evening during the first two weeks of the study; thereafter, they will receive a 265 mg tablet twice daily (BID).
  Interventions: Drug: Experimental: ALZ-801; Drug: Placebo Comparator: Placebo
- Placebo (Placebo Comparator): Subjects in the placebo treatment arm will receive placebo tablets BID throughout the study
  Interventions: Drug: Placebo Comparator: Placebo

INTERVENTIONS:
Drug: Experimental: ALZ-801 — ALZ-801 tablet 265 mg once daily in the evening for the first 2 weeks, then ALZ-801 tablet 265 mg BID
  Other Names: valiltramiprosate; tramiprosate prodrug
  Arms: ALZ-801
Drug: Placebo Comparator: Placebo — Placebo tablet BID

SUMMARY:
This study is being conducted to evaluate the safety and efficacy of ALZ-801 in Early Alzheimer's disease (AD) subjects with the APOE4/4 genotype. This is a double-blind, randomized trial with one dose of ALZ-801 compared to placebo.

DETAILED DESCRIPTION:
This is a multi-center, double-blind study that will evaluate 265 mg twice daily (BID) of ALZ-801, an oral tablet, over 78 weeks as a treatment for subjects (50-80 years old) with Early AD who are homozygous for the ε4 allele of the apolipoprotein gene (APOE4 homozygous or APOE4/4). The primary efficacy outcome assessment is a measure of cognition (ADAS-cog 13). Additional measures of global and functional impairments will also be assessed. Imaging and soluble biomarkers of AD and neurodegeneration will be measured and a sub-study to evaluate cerebrospinal fluid (CSF) biomarkers is also included.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of MCI or Mild Dementia due to AD consistent with the National Institute on Aging-Alzheimer's Association (NIA-AA) Working Group Criteria.
* Homozygous for the ε4 allele of the apolipoprotein E gene (APOE4/4).
* MMSE score at Screening of 22 to 30 (inclusive).
* CDR - Global score of 0.5 or 1 and CDR Memory Box Score of ≥ 0.5.
* RBANS delayed memory index score ≤ 85.
* Evidence of progressive memory loss over the last 12 months per investigator assessment

Exclusion Criteria:

* Brain magnetic resonance imaging (MRI) indicative of significant abnormality per central reader, other than AD related atrophy. Computed tomography (CT) scan acceptable for subjects who cannot undergo MRI.
* Diagnosis of neurodegenerative disorder other than AD.
* Diagnosis of major depressive disorder (MDD) within one year prior to screening.
* Currently taking memantine or has taken memantine within 12 weeks prior to the Baseline Visit.
* History of suicidal behavior within one year prior to screening or has ongoing suicidal ideation.
* History of seizures, excluding febrile seizures of childhood or a single distant seizure (> 5 years).
* Medically confirmed history of recent cerebral infarct or transient ischemic attack within one year prior to screening.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 325 (Actual)
Dates: Start 2021-05-19 (Actual); Primary Completion 2024-05-29 (Actual); Study Completion 2024-07-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan Abushakra, MD, Principal Investigator — Alzheon Inc.
Locations (95):
- United States (55):
  - Xenoscience, Phoenix, Arizona
  - CCT Research, Scottsdale, Arizona
  - Banner Sun Health Research Institute, Sun City, Arizona
  - ATP Clinical Research, Costa Mesa, California
  - Tilda Research, Irvine, California
  - UCSD Shiley-Marcos Alzheimer's Disease Research Center, La Jolla, California
  - Torrance Clinical Research Institute, Lomita, California
  - Collaborative NeuroScience Network LLC, Long Beach, California
  - Stanford University, Palo Alto, California
  - SC3 Research Group, Pasadena, California
  - Sutter Health, Sacramento, California
  - JEM Research Institute, Headlands Site, Atlantis, Florida
  - Bradenton Research Center, Bradenton, Florida
  - Galiz Research, Hialeah, Florida
  - Alphab Global Research, Jupiter, Florida
  - Charter Research, Lady Lake, Florida
  - K2 Medical Research, LLC, Maitland, Florida
  - Miami Jewish Health, Miami, Florida
  - Y & L Advance Health Care, Inc /DBA Elite Clinical Research, Miami, Florida
  - Mount Sinai Medical Center, Miami Beach, Florida
  - Aqualane Clinical Research, Naples, Florida
  - Charter Research, Orlando, Florida
  - Headlands Research Orlando, Orlando, Florida
  - Advanced Research Consultants, Palm Beach Gardens, Florida
  - Quantum CNS Clinical Research, Pompano Beach, Florida
  - Progressive Medical Research, Port Orange, Florida
  - ALZ Research and Treatment Center (A.R.T.C.), Stuart, Florida
  - ALZ Research and Treatment Center (A.R.T.C.), Wellington, Florida
  - Premiere Research Institute, West Palm Beach, Florida
  - Columbus Memory Center, Columbus, Georgia
  - Sandhill Research, LLC, Decatur, Georgia
  - Fort Wayne Neurological Center, Fort Wayne, Indiana
  - Louisiana State University Health Sciences Center (LSUHSC), Shreveport, Louisiana
  - Headlands Research Eastern MA, Plymouth, Massachusetts
  - WR-CRCN, Las Vegas, Nevada
  - Advanced Memory Research Center, Toms River, New Jersey
  - Neurological Associates of Albany, Albany, New York
  - NYU Alzheimer's Disease Research Center, New York, New York
  - Kline Institute for Psychiatric Research, Orangeburg, New York
  - University of Rochester Medical Center, Rochester, New York
  - Richmond Behavioral Associates, Staten Island, New York
  - Triad Clinical Trials, Greensboro, North Carolina
  - AMC Research, Matthews, North Carolina
  - NeuroScience Research Center, Canton, Ohio
  - Neurology Diagnostics, Inc., Dayton, Ohio
  - IPS Research, Oklahoma City, Oklahoma
  - Center for Cognitive Health, Portland, Oregon
  - Abington Neurological Associates, Abington, Pennsylvania
  - Lehigh Center for Clinical Research, Allentown, Pennsylvania
  - Rhode Island Mood & Memory Research Institute, East Providence, Rhode Island
  - Vanderbilt Center for Cognitive Medicine, Nashville, Tennessee
  - UT Health Science Center at Houston, Houston, Texas
  - Re:Cognition Health, Fairfax, Virginia
  - Northwest Clinical Research Center, Bellevue, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Canada (7):
  - OCT Research ULC (dba Okanagan Clinical Trials), Kelowna, British Columbia
  - Centricity Research, Halifax, Nova Scotia
  - Centricity Research, New Minas, Nova Scotia
  - Recherches Neuro-Hippocampe Inc., d/b/a Ottawa Memory Clinic, Ottawa, Ontario
  - Kawartha Centre - Redefining Healthy Aging, Peterborough, Ontario
  - Toronto Memory Program, Toronto, Ontario
  - Recherches Neuro-Hippocampe Inc. d/b/a Clinique de la Mémoire de l'Outaouais, Gatineau, Quebec
- Czechia (4):
  - Medica 111, Spol. s r.o. - Neurologicka a Rehabilitacni Ambulance Brno, Centralni Pracoviste v Brne, Brno
  - Fakultní nemocnice u sv. Anny v Brně (St. Anne's University Hospital), Brno
  - Neuropsychiatrie s.r.o., Prague
  - Vestra Clinics - Dedicated Research Clinics, Rychnov nad Kněžnou
- France (7):
  - Centre Hospitalier Universitaire de Marseille - Hôpital de la Timone, Marseille
  - Hopital Gui de Chauliac - CHRU de Montpellier, Montpellier
  - Hopital Lariboisiere - Fernand-Widal - AP-HP, Paris
  - Centre Hospitalier Universitaire (CHU) Hopitaux de Rouen, Rouen
  - Hopitaux Universitaires de Strasbourg Centre d'Investigation Clinique, Strasbourg
  - Centre de Recherche Clinique du Gerontopole - CHU Toulouse, Toulouse
  - Centre de Recherche-Hopital Geriatrique de Charpennes, Villeurbanne
- Germany (4):
  - University Hospital RWTH Aachen Neurological Study Center, Aachen
  - Klinikum der Universitaet Muenchen Innenstadt, München
  - Universitätsklinik fuer Psychiatrie und Psychotherapie, Tübingen
  - Studienzentrum Nord-West, Westerstede
- Memory Clinic, Landspitali University Hospital, Reykjavik, Iceland
- Netherlands (3):
  - Brain Research Center Den Bosch, 's-Hertogenbosch
  - Brain Research Center Amsterdam, Amsterdam
  - Brain Research Center Zwolle, Zwolle
- Spain (6):
  - Fundacia ACE - Institut Catala de Neurociencies Aplicadas, Barcelona
  - Clinica Universidad de Navarra, Madrid
  - Hospital Clinico San Carlos, Madrid
  - Clinica Universidad de Navarra, Pamplona
  - Hospital Universitari MutuaTerrassa, Terrassa
  - Centro Hospital Universitario Dr. Preset, Valencia
- United Kingdom (8):
  - Re-Cognition Health Ltd Plymouth, Plymouth, Devon
  - Re-Cognition Health Ltd London, London, Greater London
  - NeuroClin Glasgow Ltd, Motherwell, North Lanarkshire
  - Re-Cognition Health Ltd Guildford, Guildford, Surrey
  - Re-Cognition Health Ltd Birmingham, Birmingham, West Midlands
  - Re:Cognition Health Ltd Bristol, Bristol
  - St. Pancras Clinical Research, London
  - Re-Cognition Health Ltd Winchester, Winchester

REFERENCES:
- [Derived] Abushakra S, Power A, Watson D, Porsteinsson A, Sabbagh M, MacSweeney E, Cohen S, Boada Rovira M, Doraiswamy PM, Liang E, Flint S, Kesslak JP, McLaine R, Albayrak A, Schaefer J, Yu J, Tolar L, Dickson S, Hey JA, Tolar M. Clinical Efficacy, Safety and Imaging Effects of Oral Valiltramiprosate in APOEepsilon4/epsilon4 Homozygotes with Early Alzheimer's Disease: Results of the Phase III, Randomized, Double-Blind, Placebo-Controlled, 78-Week APOLLOE4 Trial. Drugs. 2025 Nov;85(11):1455-1472. doi: 10.1007/s40265-025-02250-5. Epub 2025 Sep 28. PMID 41015981

RESULTS

PARTICIPANT FLOW:
Groups:
- ALZ-801: ALZ-801 265 mg BID tablet orally. Subjects will receive placebo in the morning and one table of ALZ-801 265mg tablet in the evening during the first two weeks of the study; thereafter, they will receive a 265mg tablet BID.
  Experimental: ALZ-801: ALZ-801 tablet 265 mg BID
Period: Overall Study
Arm/Group | Placebo | ALZ-801
Started | 162 | 163
Completed | 148 | 132
Not Completed | 14 | 31
Not completed — Adverse Event | 2 | 11
Not completed — Withdrawal by Subject | 5 | 11
Not completed — Lost to Follow-up | 4 | 3
Not completed — not otherwise specified | 2 | 3
Not completed — Physician Decision | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | ALZ-801 | Total
Number analyzed (Participants) | 162 | 163 | 325
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.5 (5.93) | 68.4 (6.36) | 68.5 (6.14)
Age, Customized [Count of Participants; unit: Participants]
  50 to <=65 | 46 | 49 | 95
  >65 to 80 | 116 | 114 | 230
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 82 | 85 | 167
  Male | 80 | 78 | 158
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 2 | 3
  Black or African American | 6 | 7 | 13
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  White | 145 | 144 | 289
  Multiple Races | 1 | 1 | 2
  Race Not Reported/Missing | 9 | 9 | 18
  Hispanic/Latino | 7 | 5 | 12
  Not Hispanic/Latino | 141 | 147 | 288
  Ethnicity Not Reported | 14 | 11 | 25
Alzheimer's Diagnosis based on MMSE [Count of Participants; unit: Participants]
  Mild cognitive impairment (MCI) MMSE 27-30 | 60 | 67 | 127
  Mild Alzheimer's Disease (Mild AD) MMSE 22-26 | 102 | 96 | 198
Concomitant AChEI [Count of Participants; unit: Participants]
  Yes | 62 | 54 | 116
  No | 100 | 109 | 209
Baseline Clinical Outcomes Assessments (Safety Population) [Mean (Standard Deviation); unit: units on a scale] — The ADAS-Cog13 is a rater administered instrument with 13 items assessing areas of cognitive function most typically impaired in Alzheimer's Disease (AD). The A-IADL Questionnaire detects deficits in complex functions (activities necessary to function independently in society). CDR-SB is a semi-structured interview of participants/caregivers to rate participants' cognitive status across 6 domains of functioning. The DAD evaluates basic and instrumental activities of daily living. The MMSE is a measure of global cognition that is widely used for clinical staging of AD. Population: Not all patients had all baseline measures taken/assessed/collected at baseline.
  units on a scale
    ADAS-Cog13 | 24.31 (8.86) | 23.554 (8.26) | 23.93 (8.56)
    A-IADL-W: number analyzed (Participants) | 161 | 160 | 321
    A-IADL-W | 17.46 (20.65) | 16.00 (18.42) | 16.73 (19.55)
    CDR-SB | 2.97 (1.45) | 3.04 (1.53) | 3.00 (1.49)
    DAD: number analyzed (Participants) | 162 | 161 | 323
    DAD | 93.0 (10.34) | 93.3 (9.94) | 93.2 (10.13)
    MMSE | 25.1 (2.7) | 25.5 (2.7) | 25.3 (2.7)

OUTCOME MEASURES:

1. Primary Outcome: Primary Cognitive Efficacy Endpoint (ADAS-Cog13)
Description: Change from baseline in Alzheimer's Disease Assessment Scale - Cognitive Subscale 13 (ADAS-Cog13) scores.
  The ADAS-Cog13 is a rater administered instrument that was designed to assess the severity of the dysfunction in the cognitive and noncognitive behaviors characteristic of persons with AD. The cognitive subscale of the ADAS-Cog13 consists of 13 items assessing areas of cognitive function most typically impaired in AD: orientation, verbal memory, language, praxis, delayed free recall, digit cancellation. The ADAS-Cog13 scale ranges from 0 to 85. Higher scores indicate greater disease severity.
Time Frame: Baseline to Week 78
Population: Full Analysis Set (FAS): The FAS includes all study subjects who received at least one dose of the study drug, had at least one baseline assessment and any post baseline efficacy assessment. All primary and secondary clinical efficacy analyses are conducted on this population.
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Placebo | ALZ-801
Number analyzed (Participants) | 158 | 162
Score on a scale | 4.40 (0.69) | 3.89 (0.69)
Statistical Analysis 1: Comparison: Placebo vs ALZ-801; The null hypothesis was change from baseline (CBL) of ADAS-Cog13 in the ALZ-801 arm was not different from the placebo arm. The alternative hypothesis was that the CBL of ADAS-Cog13 in ALZ-801 arm was different. A Mixed-Effect Model Repeated Measure (MMRM) model was used with fixed terms for treatment, gender, age group, disease severity based on baseline MMSE (≤ 26 vs. > 26), concomitant AD medications, visit, and treatment by visit interaction and baseline ADAS-Cog 13 values as covariates; Test type: Other — For the primary efficacy outcome of ADAS-Cog 13, this study has >90% power to detect a 3.0-point difference between the active ALZ-801 treatment and the placebo in the CBL to Week 78. An increase in ADAS-Cog scores denotes cognitive worsening. The primary analysis population was the full analysis set (FAS). The FAS included all study subjects who received at least one dose of the study drug and had at least one baseline assessment and any post baseline efficacy assessment; p = 0.6058, MMRM — Statistical testing was two-sided at the α=0.05 significance level. Between-treatment group comparison (effect in ALZ-801 minus effect in placebo): LSM difference and p-value; Least Squares Mean Difference = -0.51, Standard Error of Mean 0.98 — ALZ-801 minus placebo

2. Primary Outcome: Incidence, Nature, and Severity of Treatment Emergent Adverse Events (TEAE)
Description: Safety and tolerability as measured by incidence, nature and severity of treatment emergent adverse events (TEAE), serious TEAEs, and TEAEs leading to withdrawal.
Time Frame: Entire study: approximately 82 weeks. (first dose of study drug until end of Safety Follow-up Visit at 28 +/- 7 days after the last dose (ie, 78-week treatment period plus 4-weeks follow-up after last dose up to total of 82 weeks)
Population: Safety Population: subjects who took at least 1 dose of any study drug are included.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | ALZ-801
Number analyzed (Participants) | 162 | 163
Participants
  TEAE | 137 | 140
  Study drug related TEAE | 44 | 75
  Serious TEAE | 13 | 14
  Serious study drug related TEAE | 0 | 1
  TEAE leading to discontinuation of study drug | 4 | 13
  Study drug related TEAE leading to study drug discontinuation | 1 | 10

3. Secondary Outcome: Key Secondary Endpoint (A-IADL-W)
Description: Change from baseline in Amsterdam - Instrumental Activities of Daily Living scores calculated using the weighted average method (A-IADL-W score). The A-IADL Questionnaire is a 70-item informant-based computerized questionnaire aimed at detecting deficits in complex functions at the early stages of AD. Instrumental ADL can be described as the activities necessary to function independently in society. These activities include, but are not limited to, cooking, doing finances, and shopping. They are complex everyday tasks, determined by multiple cognitive processes and controlled processing. They can be distinguished from basic ADL, which include basic self-care skills. The A-IADL-W has a score range of 0-100 and is calculated as follows: (sum of all scores / number of questions scored) × 25. For A-IADL-W, higher scores indicates worse functioning or more impairment.
Time Frame: Baseline to Week 78
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | ALZ-801
Number analyzed (Participants) | 158 | 162
score on a scale | 13.59 (2.02) | 13.60 (2.00)
Statistical Analysis 1: Comparison: Placebo vs ALZ-801; The A-IADL-W is one of 2 key secondary endpoints. The key secondary efficacy endpoints were to be compared only after the comparison of the primary endpoint has reached statistical significance. Because the primary endpoint did not reach statistical significance, the comparisons for the key secondary endpoints are descriptive only. The same MMRM method applied to the primary efficacy endpoint was used to evaluate the between-treatment difference for the key secondary endpoints; Test type: Other; p = 0.9966, MMRM — Nominal p-value; Nominal (descriptive only); Least Squares Mean Difference = 0.01, Standard Error of Mean 2.84 — ALZ-801 minus placebo

4. Secondary Outcome: Key Secondary Endpoint (CDR-SB)
Description: Change from baseline in Clinical Dementia Rating - Sum of Boxes (CDR-SB) scores. CDR-SB is a semi-structured interview of participants and their caregivers. Participant's cognitive status is rated across 6 domains of functioning, including memory, orientation, judgment/problem solving, community affairs, home/hobbies, and personal care. Severity score assigned for each of 6 domains; Total score (SB) ranges from 0 to 18. Higher scores indicate greater disease severity.
Time Frame: Baseline to Week 78
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | ALZ-801
Number analyzed (Participants) | 158 | 162
score on a scale | 1.36 (0.21) | 1.05 (0.22)
Statistical Analysis 1: Comparison: Placebo vs ALZ-801; The CDR-SB is one of 2 key secondary endpoints. The key secondary efficacy endpoints were to be compared only after the comparison of the primary endpoint has reached statistical significance. Because the primary endpoint did not reach statistical significance, the comparisons for the key secondary endpoints are descriptive only. The same MMRM method applied to the primary efficacy endpoint was used to evaluate the between-treatment difference for the key secondary endpoints; Test type: Other; p = 0.3090, MMRM — Nominal p-value; Least Squares Mean Difference = -0.31, Standard Error of Mean 0.31 — ALZ-801 minus placebo

5. Secondary Outcome: Functional Assessment (DAD)
Description: Change from baseline in Disability Assessment for Dementia (DAD)scores. The DAD consists of 40 items with a score range of 0-100 to evaluate the basic and instrumental activities of daily living of subjects with dementia. It is administered through an interview with the caregiver. Higher DAD scores indicate less disability or better function.
Time Frame: Baseline to Week 78
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | ALZ-801
Number analyzed (Participants) | 158 | 162
score on a scale | -9.2 (1.7) | -6.5 (1.7)
Statistical Analysis 1: Comparison: Placebo vs ALZ-801; The same MMRM method applied to the primary efficacy endpoint was used to evaluate the between-treatment difference for the additional secondary endpoints. The hypothesis testing was done without control for type I errors due to multiple comparisons, and the p-value was considered nominal; Test type: Other; p = 0.2763, MMRM — Nominal p-value; Nominal (descriptive only); Least Squares Mean Difference = 2.6, Standard Error of Mean 2.4 — ALZ-801 minus placebo

6. Secondary Outcome: Global Cognition Assessment (MMSE)
Description: Change from baseline in Mini-Mental State Examination (MMSE) score. The MMSE is a measure of global cognition that is widely used for clinical staging of Alzheimer's Disease. It consists of 11 domains items for a score range of 0-30 to assess general cognitive function. Higher score on MMSE means better cognitive skills.
Time Frame: Baseline to Week 78
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | ALZ-801
Number analyzed (Participants) | 158 | 162
score on a scale | -2.03 (0.33) | -1.60 (0.33)
Statistical Analysis 1: Comparison: Placebo vs ALZ-801; [analysis description as in outcome 5, analysis 1]; Test type: Other; p = 0.4484, MMRM — Nominal p-value; Nominal (descriptive only); Least Squares Mean Difference = 0.35, Standard Error of Mean 0.47 — ALZ-801 minus placebo

7. Other Pre Specified Outcome: Imaging Biomarker Endpoint (Hippocampal Volume)
Description: Change from baseline in total (bilateral) hippocampal volume (HV) (uL) as measured by Magnetic Resonance Imaging (MRI). HV atrophy is an early event in AD patients, especially in APOE4/4 homozygotes who show accelerated atrophy compared to APOE3/3 patients with Early AD. HV may be a marker of synaptic loss and neurodegeneration.
Time Frame: Baseline to Week 78
Population: The Imaging Biomarker population included all subjects with an evaluable baseline vMRI assessment who had received at least 1 dose of study drug and had at least 1 evaluable post-baseline imaging vMRI assessment.
Measure: Least Squares Mean (Standard Error); unit: microliters
Arm/Group | Placebo | ALZ-801
Number analyzed (Participants) | 144 | 146
microliters | -418.5 (21.46) | -345.0 (22.01)
Statistical Analysis 1: Comparison: Placebo vs ALZ-801; Analysis of the volumetric MRI outcomes were performed using the same MMRM approach described for analysis of the primary clinical endpoint. The MMRM model included treatment, the use of concomitant AD medications (AChEI or none), age group (50 through 65 years or > 65 years), gender, disease severity based on baseline MMSE, baseline volumetric MRI value, visit, and treatment by visit interaction. The MRI magnet strength (1.5 or 3 Tesla) was also included as a covariate in the model; Test type: Other; p = 0.0174, MMRM — Nominal p-value; Least Squares Mean Difference = 73.505, Standard Error of Mean 30.711 — ALZ-801 minus placebo

8. Other Pre Specified Outcome: Imaging Biomarker Endpoint (Cortical Thickness [Whole Cortex])
Description: Change from baseline in total (bilateral) cortical thickness (mm) as measured by MRI. Brain MRI studies in Alzheimer's Disease patients show progressive cortical atrophy, reflecting progressive neurodegeneration.
Time Frame: Baseline to Week 78
Population: Imaging Biomarker Population
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | Placebo | ALZ-801
Number analyzed (Participants) | 144 | 146
mm | -0.060 (0.003) | -0.048 (0.003)
Statistical Analysis 1: Comparison: Placebo vs ALZ-801; [analysis description as in outcome 7, analysis 1]; Test type: Other; p = 0.0020, MMRM — Nominal p-value; Least Squares Mean Difference = 0.012, Standard Error of Mean 0.004 — ALZ-801 minus placebo

9. Other Pre Specified Outcome: Imaging Biomarker Endpoint (Cortical Thickness [Mayo Index])
Description: Change from baseline in total (bilateral) cortical thickness (mm) as measured by MRI. Brain MRI studies in Alzheimer's Disease patients show progressive cortical atrophy, reflecting progressive neurodegeneration. The Mayo Index refers specifically to the measurement of cortical thickness in the medial temporal lobe.
Time Frame: Baseline to Week 78
Population: Imaging Biomarker Population
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | Placebo | ALZ-801
Number analyzed (Participants) | 144 | 146
mm | -0.121 (0.005) | -0.099 (0.005)
Statistical Analysis 1: Comparison: Placebo vs ALZ-801; [analysis description as in outcome 7, analysis 1]; Test type: Other; p = 0.0040, MMRM — Nominal p-value; Least Squares Mean Difference = 0.021, Standard Error of Mean 0.007 — ALZ-801 minus placebo

10. Other Pre Specified Outcome: Imaging Biomarker Endpoint (Whole Brain Volume)
Description: Change from baseline in whole brain volume (uL) as measured by Magnetic Resonance Imaging (MRI).
Time Frame: Baseline to Week 78
Population: Imaging Biomarker Population
Measure: Least Squares Mean (Standard Error); unit: microliters
Arm/Group | Placebo | ALZ-801
Number analyzed (Participants) | 144 | 146
microliters | -17877.0 (955.98) | -15056.0 (979.86)
Statistical Analysis 1: Comparison: Placebo vs ALZ-801; [analysis description as in outcome 7, analysis 1]; Test type: Other; p = 0.0400, MMRM — Nominal p-value; Least Squares Mean Difference = 2821.027, Standard Error of Mean 1366.533 — ALZ-801 minus placebo

11. Other Pre Specified Outcome: Imaging Biomarker Endpoint (Ventricular Volume)
Description: Change from baseline in total (bilateral) ventricular volume (uL) as measured by Magnetic Resonance Imaging (MRI).
Time Frame: Baseline to Week 78
Population: Imaging Biomarker Population
Measure: Least Squares Mean (Standard Error); unit: microliters
Arm/Group | Placebo | ALZ-801
Number analyzed (Participants) | 144 | 146
microliters | 5186.3 (256.19) | 4028.9 (262.86)
Statistical Analysis 1: Comparison: Placebo vs ALZ-801; Test type: Other; p = 0.0018, MMRM — Nominal p-value; Least Squares Mean Difference = -1157, Standard Error of Mean 367

12. Other Pre Specified Outcome: Imaging Biomarker Endpoint - DTI in Grey Matter Mean Diffusivity - Bilateral Caudate
Description: Change from baseline in Grey Matter Mean Diffusivity (Bilateral Caudate) as measured by Diffusion Tensor Imaging - Magnetic Resonance Imaging (DTI-MRI). The mean diffusivity (MD) is the average of the three main diffusion values (eigenvalues) obtained from the diffusion tensor imaging (DTI). It is expressed as mm2/s. This unit quantifies the average rate of water diffusion across all directions within a tissue, providing an overall measure of tissue microstructural properties. Lower MD value suggests better maintenance of microstructural integrity of a given brain tissue. Positive treatment effects of ALZ-801 on DTI would present as lower mean diffusivity compared with the placebo group.
Time Frame: Baseline to Week 78
Population: DTI-MRI Population defined as all participants who had an evaluable baseline DTI-MRI assessment, received at least one dose of study drug, and had at least one evaluable post-baseline DTI-MRI assessment.
Measure: Least Squares Mean (Standard Error); unit: square millimeters per second (mm²/s)
Arm/Group | Placebo | ALZ-801
Number analyzed (Participants) | 103 | 105
square millimeters per second (mm²/s) | 0.000028 (0.00000775) | 0.000007439 (0.00000792)
Statistical Analysis 1: Comparison: Placebo vs ALZ-801; Analysis of the DTI-MRI outcomes were performed using the same MMRM approach described for analysis of the primary clinical endpoint. The MMRM model included treatment, the use of concomitant AD medications (AChEI or none), age group (50 through 65 years or > 65 years), gender, disease severity based on baseline MMSE, baseline DTI-MRI value, visit, and treatment by visit interaction. The MRI magnet strength (1.5 or 3 Tesla) was also included as a covariate in the model; Test type: Other; p = 0.054, MMRM — Nominal p-value; Least Squares Mean Difference = -0.0000214, 95% CI 2-sided [-0.0000432 to 0.00000037], Standard Error of Mean 0.00000111 — ALZ-801 minus placebo

13. Other Pre Specified Outcome: Imaging Biomarker Endpoint - DTI in White Matter Mean Diffusivity (Bilateral Fornix)
Description: Change from baseline in Bilateral Fornix White Matter Mean Diffusivity as measured by Diffusion Tensor Imaging - Magnetic Resonance Imaging (DTI-MRI). The mean diffusivity (MD) is the average of the three main diffusion values (eigenvalues) obtained from the diffusion tensor imaging (DTI). It is expressed as mm2/s. This unit quantifies the average rate of water diffusion across all directions within a tissue, providing an overall measure of tissue microstructural properties. Lower MD value suggests better maintenance of microstructural integrity of a given brain tissue. Positive treatment effects of ALZ-801 on DTI would present as lower mean diffusivity compared with the placebo group.
Time Frame: Baseline to Week 78
Population: DTI-MRI Population
Measure: Least Squares Mean (Standard Error); unit: square millimeters per second (mm²/s)
Arm/Group | Placebo | ALZ-801
Number analyzed (Participants) | 103 | 105
square millimeters per second (mm²/s) | 0.0000237 (0.0000058) | 0.000000843 (0.00000593)
Statistical Analysis 1: Comparison: Placebo vs ALZ-801; Test type: Other; p = 0.0064, MMRM — Nominal p-value; Least Squares Mean Difference = -0.0000228, 95% CI 2-sided [-0.0000391 to -0.0000065], Standard Error of Mean 0.00000829

14. Other Pre Specified Outcome: Imaging Biomarker Endpoint - White Matter Fractional Anisotropy (Bilateral Fornix)
Description: Change from baseline in Bilateral Fornix White Matter Fractional Anisotropy as measured by Diffusion Tensor Imaging - Magnetic Resonance Imaging (DTI-MRI). Fractional anisotropy (FA) is a unitless, scalar value that measures the degree of anisotropic (directional) water diffusion within a voxel, ranging from 0 to 1. A value of 0 indicates perfectly isotropic (equal in all directions) diffusion, while a value of 1 indicates perfectly anisotropic (directional) diffusion. Higher FA value suggests better maintenance of microstructural integrity of a given brain tissue. Positive treatment effects of ALZ-801 on DTI would present as higher FA in the ALZ-801 group compared with the placebo group.
Time Frame: Baseline to Week 78
Population: DTI-MRI Population
Measure: Least Squares Mean (Standard Error); unit: Units on a scale (fractions 0-1)
Arm/Group | Placebo | ALZ-801
Number analyzed (Participants) | 103 | 105
Units on a scale (fractions 0-1) | -0.0154 (0.00332) | -0.002089 (0.00336)
Statistical Analysis 1: Comparison: Placebo vs ALZ-801; Test type: Other; p = 0.0465, MMRM — Nominal p-value; Least Squares Mean Difference = 0.009455, 95% CI 2-sided [0.0001469 to 0.01876], Standard Error of Mean 0.00472

15. Other Pre Specified Outcome: Cognitive Efficacy Endpoint (ADAS-Cog 13) - MCI Subgroup
Description: Change from baseline in Alzheimer's Disease Assessment Scale - Cognitive Subscale 13 (ADAS-cog 13) scores at 78 weeks.
  The ADAS-Cog13 is a rater administered instrument that was designed to assess the severity of the dysfunction in the cognitive and noncognitive behaviors characteristic of persons with AD. The cognitive subscale of the ADAS-Cog13 consists of 13 items assessing areas of cognitive function most typically impaired in AD: orientation, verbal memory, language, praxis, delayed free recall, digit cancellation. The ADAS-Cog13 scale ranges from 0 to 85. Higher scores indicate greater disease severity.
Time Frame: Baseline to Week 78
Population: FAS MCI subgroup: all study subjects in the MCI subgroup who received at least one dose of the study drug, had at least one baseline assessment and any post baseline efficacy assessment.
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Placebo | ALZ-801
Number analyzed (Participants) | 58 | 67
Score on a scale | 4.10 (0.81) | 1.97 (0.83)
Statistical Analysis 1: Comparison: Placebo vs ALZ-801; Test type: Other; p = 0.0416, MMRM — Nominal p-value; Least Squares Mean Difference = -2.14, Standard Error of Mean 1.05

16. Other Pre Specified Outcome: Cognitive Efficacy Endpoint (ADAS-Cog 13) - Mild Alzheimer's Disease(Mild AD) Subgroup
Description: as for outcome 15
Time Frame: Baseline to Week 78
Population: FAS Mild AD subgroup: all study subjects in the Mild AD subgroup who received at least one dose of the study drug, had at least one baseline assessment and any post baseline efficacy assessment.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | ALZ-801
Number analyzed (Participants) | 100 | 95
score on a scale | 4.79 (0.75) | 5.66 (0.75)
Statistical Analysis 1: Comparison: Placebo vs ALZ-801; Test type: Other; p = 0.3945, MMRM — Nominal p-value; Least Squares Mean Difference = 0.87, Standard Error of Mean 1.02

17. Other Pre Specified Outcome: A-IADL-W - MCI Subgroup
Description: as for outcome 3
Time Frame: Baseline to Week 78
Population: FAS MCI Subgroup
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | ALZ-801
Number analyzed (Participants) | 58 | 67
score on a scale | 4.84 (2.45) | 1.43 (2.50)
Statistical Analysis 1: Comparison: Placebo vs ALZ-801; Test type: Other; p = 0.2682, MMRM — Nominal p-value; Least Squares Mean Difference = -3.41, Standard Error of Mean 3.07

18. Other Pre Specified Outcome: A-IADL-W - Mild AD Subgroup
Description: as for outcome 3
Time Frame: Baseline to Week 78
Population: FAS Mild AD Subgroup
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | ALZ-801
Number analyzed (Participants) | 100 | 95
score on a scale | 18.55 (2.21) | 22.20 (2.21)
Statistical Analysis 1: Comparison: Placebo vs ALZ-801; Test type: Other; p = 0.2178, MMRM — Nominal p-value; Least Squares Mean Difference = 3.66, Standard Error of Mean 2.96

19. Other Pre Specified Outcome: CDR-SB - MCI Subgroup
Description: as for outcome 4
Time Frame: Baseline to Week 78
Population: FAS MCI Subgroup
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | ALZ-801
Number analyzed (Participants) | 58 | 67
score on a scale | 0.63 (0.26) | -0.02 (0.27)
Statistical Analysis 1: Comparison: Placebo vs ALZ-801; Test type: Other; p = 0.0533, MMRM — Nominal p-value; Least Squares Mean Difference = -0.646, Standard Error of Mean 0.333

20. Other Pre Specified Outcome: CDR-SB - Mild AD Subgroup
Description: as for outcome 4
Time Frame: Baseline to Week 78
Population: FAS Mild AD Subgroup
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | ALZ-801
Number analyzed (Participants) | 100 | 95
score on a scale | 1.84 (0.23) | 1.97 (0.24)
Statistical Analysis 1: Comparison: Placebo vs ALZ-801; Test type: Other; p = 0.6854, MMRM — Nominal p-value; Least Squares Mean Difference = 0.127, Standard Error of Mean 0.314

21. Other Pre Specified Outcome: Functional Assessment (DAD) - MCI Subgroup
Description: as for outcome 5
Time Frame: Baseline to Week 78
Population: FAS MCI Subgroup
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | ALZ-801
Number analyzed (Participants) | 58 | 67
score on a scale | -6.3 (1.9) | -0.2 (2.0)
Statistical Analysis 1: Comparison: Placebo vs ALZ-801; Test type: Other; p = 0.0161, MMRM — Nominal p-value; Least Squares Mean Difference = 6.10, Standard Error of Mean 2.52

22. Other Pre Specified Outcome: Functional Assessment (DAD) - Mild AD Subgroup
Description: as for outcome 5
Time Frame: Baseline to Week 78
Population: FAS Mild AD Subgroup
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | ALZ-801
Number analyzed (Participants) | 100 | 95
score on a scale | -11.1 (1.8) | -11.6 (1.8)
Statistical Analysis 1: Comparison: Placebo vs ALZ-801; Test type: Other; p = 0.8387, MMRM — Nominal p-value; Least Squares Mean Difference = -0.51, Standard Error of Mean 2.51

23. Other Pre Specified Outcome: Global Cognition Assessment (MMSE) - MCI Subgroup
Description: as for outcome 6
Time Frame: Baseline to Week 78
Population: FAS MCI Subgroup
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Placebo | ALZ-801
Number analyzed (Participants) | 58 | 67
Score on a scale | -1.4 (0.4) | -0.5 (0.4)
Statistical Analysis 1: Comparison: Placebo vs ALZ-801; Test type: Other; p = 0.0795, MMRM — Nominal p-value; Least Squares Mean Difference = 0.9, 95% CI 2-sided [-0.103 to 1.845], Standard Error of Mean 0.5

24. Other Pre Specified Outcome: Global Cognition Assessment (MMSE) - Mild AD Subgroup
Description: as for outcome 6
Time Frame: Baseline to Week 78
Population: FAS Mild AD Subgroup
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | ALZ-801
Number analyzed (Participants) | 100 | 95
score on a scale | -2.6 (0.4) | -2.7 (0.4)
Statistical Analysis 1: Comparison: Placebo vs ALZ-801; Test type: Other; p = 0.8169, MMRM — Nominal p-value; Least Squares Mean Difference = -0.1, 95% CI 2-sided [-1.070 to 0.845], Standard Error of Mean 0.5

25. Other Pre Specified Outcome: Hippocampal Volume (MCI Subgroup)
Description: as for outcome 7
Time Frame: Baseline to Week 78
Population: Imaging Biomarker Population MCI Subgroup: this population included all subjects in the MCI subgroup with an evaluable baseline vMRI assessment who had received at least 1 dose of study drug and had at least 1 evaluable post-baseline imaging vMRI assessment.
Measure: Least Squares Mean (Standard Error); unit: microliters
Arm/Group | Placebo | ALZ-801
Number analyzed (Participants) | 52 | 61
microliters | -411.2 (29.60) | -303.1 (30.16)
Statistical Analysis 1: Comparison: Placebo vs ALZ-801; Test type: Other; p = 0.0042, MMRM — Nominal p-value; Least Squares Mean Difference = 108.1, Standard Error of Mean 37.46

26. Other Pre Specified Outcome: Hippocampal Volume (Mild AD Subgroup)
Description: as for outcome 7
Time Frame: Baseline to Week 78
Population: Imaging Biomarker Population Mild AD Subgroup: this population included all subjects with an evaluable baseline vMRI assessment who had received at least 1 dose of study drug and had at least 1 evaluable post-baseline imaging vMRI assessment.
Measure: Least Squares Mean (Standard Error); unit: microliters
Arm/Group | Placebo | ALZ-801
Number analyzed (Participants) | 92 | 85
microliters | -423.2 (23.27) | -371.8 (24.75)
Statistical Analysis 1: Comparison: Placebo vs ALZ-801; Test type: Other; p = 0.1145, MMRM — Nominal p-value; Least Squares Mean Difference = 51.3, Standard Error of Mean 32.42

27. Other Pre Specified Outcome: Cortical Thickness (Whole Cortex) (MCI Subgroup)
Description: as for outcome 8
Time Frame: Baseline to Week 78
Population: Imaging Biomarker Population MCI Subgroup
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | Placebo | ALZ-801
Number analyzed (Participants) | 52 | 61
mm | -0.059 (0.004) | -0.038 (0.004)
Statistical Analysis 1: Comparison: Placebo vs ALZ-801; Test type: Other; p < 0.0001, MMRM — Nominal p-value; Least Squares Mean Difference = 0.020, Standard Error of Mean 0.005

28. Other Pre Specified Outcome: Cortical Thickness (Whole Cortex) (Mild AD Subgroup)
Description: as for outcome 8
Time Frame: Baseline to Week 78
Population: Imaging Biomarker Population Mild AD Subgroup
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | Placebo | ALZ-801
Number analyzed (Participants) | 92 | 85
mm | -0.061 (0.003) | -0.054 (0.003)
Statistical Analysis 1: Comparison: Placebo vs ALZ-801; Test type: Other; p = 0.0985, MMRM — Nominal p-value; Least Squares Mean Difference = 0.007, Standard Error of Mean 0.004

29. Other Pre Specified Outcome: Cortical Thickness (Mayo Index) (MCI Subgroup)
Description: Change from baseline in total (bilateral) cortical thickness (mm) as measured by MRI. Brain MRI studies in Alzheimer's Disease patients show progressive cortical atrophy, reflecting progressive neurodegeneration. The Mayo Index refers specifically to the measurement of cortical thickness in the medial temporal lobe versus the whole cortex.
Time Frame: Baseline to Week 78
Population: Imaging Biomarker Population MCI Subgroup
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | Placebo | ALZ-801
Number analyzed (Participants) | 52 | 61
mm | -0.117 (0.007) | -0.084 (0.007)
Statistical Analysis 1: Comparison: Placebo vs ALZ-801; Test type: Other; p = 0.0002, MMRM — Nominal p-value; Least Squares Mean Difference = 0.033, Standard Error of Mean 0.009

30. Other Pre Specified Outcome: Cortical Thickness (Mayo Index) (Mild AD Subgroup)
Description: as for outcome 29
Time Frame: Baseline to Week 78
Population: Imaging Biomarker Population Mild AD Subgroup
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | Placebo | ALZ-801
Number analyzed (Participants) | 92 | 85
mm | -0.123 (0.006) | -0.109 (0.006)
Statistical Analysis 1: Comparison: Placebo vs ALZ-801; Test type: Other; p = 0.0699, MMRM — Nominal p-value; Least Squares Mean Difference = 0.014, Standard Error of Mean 0.008

31. Other Pre Specified Outcome: Whole Brain Volume (MCI Subgroup)
Description: Change from baseline in whole brain volume (uL) as measured by Magnetic Resonance Imaging (MRI).
Time Frame: Baseline to Week 78
Population: Imaging Biomarker Population MCI Subgroup
Measure: Least Squares Mean (Standard Error); unit: microliters
Arm/Group | Placebo | ALZ-801
Number analyzed (Participants) | 52 | 61
microliters | -17559.5 (1417.91) | -13715.7 (1449.14)
Statistical Analysis 1: Comparison: Placebo vs ALZ-801; Test type: Other; p = 0.0267, MMRM — Nominal p-value; Least Squares Mean Difference = 3843.824, Standard Error of Mean 1726.729

32. Other Pre Specified Outcome: Whole Brain Volume (Mild AD Subgroup)
Description: Change from baseline in whole brain volume (uL) as measured by Magnetic Resonance Imaging (MRI).
Time Frame: Baseline to Week 78
Population: Imaging Biomarker Population Mild AD Subgroup
Measure: Least Squares Mean (Standard Error); unit: microliters
Arm/Group | Placebo | ALZ-801
Number analyzed (Participants) | 92 | 85
microliters | -18081.4 (1056.74) | -15917.1 (1143.24)
Statistical Analysis 1: Comparison: Placebo vs ALZ-801; Test type: Other; p = 0.1386, MMRM — Nominal p-value; Least Squares Mean Difference = 2164.299, Standard Error of Mean 1457.282

33. Other Pre Specified Outcome: Ventricular Volume (MCI Subgroup)
Description: Change from baseline in total (bilateral) ventricular volume (uL) as measured by Magnetic Resonance Imaging (MRI).
Time Frame: Baseline to Week 78
Population: Imaging Biomarker Population MCI Subgroup
Measure: Least Squares Mean (Standard Error); unit: microliters
Arm/Group | Placebo | ALZ-801
Number analyzed (Participants) | 52 | 61
microliters | 4490.5 (343.65) | 3178.2 (350.44)
Statistical Analysis 1: Comparison: Placebo vs ALZ-801; Test type: Other; p = 0.0029, MMRM — Nominal p-value; Least Squares Mean Difference = -1312, Standard Error of Mean 437

34. Other Pre Specified Outcome: Ventricular Volume (Mild AD Subgroup)
Description: Change from baseline in total (bilateral) ventricular volume (uL) as measured by Magnetic Resonance Imaging (MRI).
Time Frame: Baseline to Week 78
Population: Imaging Biomarker Population Mild AD Subgroup
Measure: Least Squares Mean (Standard Error); unit: microliters
Arm/Group | Placebo | ALZ-801
Number analyzed (Participants) | 92 | 85
microliters | 5630.4 (274.91) | 4573.4 (294.71)
Statistical Analysis 1: Comparison: Placebo vs ALZ-801; Test type: Other; p = 0.0065, MMRM — Nominal p-value; Least Squares Mean Difference = -1057, Standard Error of Mean 386

35. Post Hoc Outcome: Cerebellar Volume
Description: Change from baseline in total (bilateral) cerebellar volume (uL) as measured by Magnetic Resonance Imaging (MRI).
Time Frame: Baseline to Week 78
Population: Imaging Biomarker Population
Measure: Least Squares Mean (Standard Error); unit: microliters
Arm/Group | Placebo | ALZ-801
Number analyzed (Participants) | 144 | 146
microliters | -577.0 (62.50) | -427.2 (64.70)
Statistical Analysis 1: Comparison: Placebo vs ALZ-801; [analysis description as in outcome 7, analysis 1]; Test type: Other; p = 0.0966, MMRM — Nominal p-value; Least Squares Mean Difference = 149.800, Standard Error of Mean 89.801

36. Post Hoc Outcome: Cerebellar Volume (MCI Subgroup)
Description: Change from baseline in total (bilateral) cerebellar volume (uL) as measured by Magnetic Resonance Imaging (MRI).
Time Frame: Baseline to Week 78
Population: Imaging Biomarker Population MCI Subgroup
Measure: Least Squares Mean (Standard Error); unit: microliters
Arm/Group | Placebo | ALZ-801
Number analyzed (Participants) | 52 | 61
microliters | -566.8 (91.78) | -428.8 (94.09)
Statistical Analysis 1: Comparison: Placebo vs ALZ-801; Test type: Other; p = 0.2200, MMRM — Nominal p-value; Least Squares Mean Difference = 137.943, Standard Error of Mean 112.257

37. Post Hoc Outcome: Cerebellar Volume (Mild AD Subgroup)
Description: Change from baseline in total (bilateral) cerebellar volume (uL) as measured by Magnetic Resonance Imaging (MRI).
Time Frame: Baseline to Week 78
Population: Imaging Biomarker Population Mild AD Subgroup
Measure: Least Squares Mean (Standard Error); unit: microliters
Arm/Group | Placebo | ALZ-801
Number analyzed (Participants) | 92 | 85
microliters | -583.6 (68.62) | -426.2 (75.18)
Statistical Analysis 1: Comparison: Placebo vs ALZ-801; Test type: Other; p = 0.1005, MMRM — Nominal p-value; Least Squares Mean Difference = 157.414, Standard Error of Mean 95.523

ADVERSE EVENTS:
Time Frame: All AEs (deaths, Serious Adverse Events, Other Adverse Events) were recorded for up to 95 weeks (13 weeks screening + 78-week treatment + 4 weeks follow-up). All AEs were collected from ICF signing at screening through Safety Follow-up Visit 4 weeks after last efficacy visit at week 78. Medical conditions present at screening were captured as medical history. However, if a condition deteriorated, it was recorded as an AE.
Arm/Group | Placebo | ALZ-801
All-Cause Mortality (participants affected / at risk) | 0/162 | 0/163
Serious Adverse Events (participants affected / at risk) | 13/162 | 15/163
Other Adverse Events (participants affected / at risk) | 94/162 | 104/163
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=162) | ALZ-801 (N=163)
Angina Pectoris (Cardiac disorders) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac Failure (Cardiac disorders) | 0 (0) | 1 (1)
Coronary Artery Stenosis (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial Infarction (Cardiac disorders) | 1 (1) | 1 (1)
Myocardial Injury (Cardiac disorders) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 1 (1)
Intestinal Obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Chest Pain (General disorders) | 1 (1) | 0 (0)
Cholecystitis Acute (Hepatobiliary disorders) | 0 (0) | 1 (1)
Gallbladder necrosis (Hepatobiliary disorders) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 1 (1) | 0 (0)
Cholecystitis Infective (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia Aspiration (Infections and infestations) | 0 (0) | 1 (1)
Pyelonephritis Acute (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Ankle Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Bladder Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Femur Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Incarcerated Incisional Hernia (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Pelvic Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Blood Calcium Increased (Investigations) | 0 (0) | 1 (1)
Blood Potassium Decreased (Investigations) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Malignant Melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Thyroid Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cerebrovascular Accident (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 2 (2)
Transient Ischaemic Attack (Nervous system disorders) | 1 (1) | 0 (0)
Paranoia (Psychiatric disorders) | 0 (0) | 1 (2)
Psychotic Disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Renal Colic (Renal and urinary disorders) | 1 (1) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=162) | ALZ-801 (N=163)
COVID-19 (Infections and infestations) | 33 | 35
Nausea (Gastrointestinal disorders) | 8 | 42
Weight Decreased (Investigations) | 12 | 23
Fall (Injury, poisoning and procedural complications) | 11 | 10
Headache (Nervous system disorders) | 13 | 9
Urinary Tract Infection (Infections and infestations) | 13 | 10
Cerebral Microhaemorrhage (Nervous system disorders) | 12 | 8
Decreased Appetite (Metabolism and nutrition disorders) | 3 | 16
Dizziness (Nervous system disorders) | 9 | 9
Vomiting (Gastrointestinal disorders) | 2 | 16
Amyloid related imaging abnormality - microhaemorrhages and heamosiderin deposits (Nervous system disorders) | 9 | 6
Anxiety (Psychiatric disorders) | 9 | 6
Back pain (Musculoskeletal and connective tissue disorders) | 11 | 5
Hypertension (Vascular disorders) | 9 | 7
Diarrhoea (Gastrointestinal disorders) | 9 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2022-01-24): https://cdn.clinicaltrials.gov/large-docs/20/NCT04770220/Prot_000.pdf
  • Statistical Analysis Plan (2024-04-04): https://cdn.clinicaltrials.gov/large-docs/20/NCT04770220/SAP_001.pdf